CLINICAL TRIAL: NCT03113734
Title: Construction and Validation of a Functional Score for the Detection of Ruptures of the Anterior Cruciate Ligament in the Immediate Post-traumatic Period
Brief Title: Clinical Screening of Acute Ruptures of the Anterior Cruciate Ligament of the Knee
Acronym: ACL-TS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: French Arthroscopic Society (Other)
Collaborators: Fondation Paul Bennetot (Other); Clinique les Maussins (Unknown); Clinique Mutualiste de Lorient (Unknown)
Responsible Party: Sponsor
Other Study IDs: SFA-ACL-TS 2015
Record Dates: First submitted 2017-04-09; First posted 2017-04-14 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Orthopedic; Rupture
MeSH Terms: conditions — Rupture | interventions — Facility Design and Construction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Construction and validation of a functional score — All patients will be treated at the same way:
  Completion of questionnaire by the physician with him. Once the consultation has been completed, the physician will issue prescriptions for the usual medical treatment, laximetry prescription (GNRB) to be performed when the knee is indolent and the prescription of the MRI to be performed .The physician will inform the patient that they should consult with the investigator's orthopedic surgeon once the results of GNRB and MRI are available.The study will end there for the patient. The surgeon will then follow his usual diagnostic procedure to decide on the future care of the patient.

SUMMARY:
This study develops the construction and validation of a reliable functional screening score in LCA ruptures in the immediate post-traumatic period.

This score, realizable in an emergency, would be an early warning signal requiring an emergency consultation with an orthopedic surgeon. It would be a tool for screening acute LCA ruptures at a time when ligament testing maneuvers are too painful to be contributory to the diagnosis. It would avoid a premature return to dangerous activity for the knee with a rupture of the LCA.

The other impact would be economical since it would avoid the realization of unnecessary MRI.

On the other hand, it will allow patients with LCA rupture to have faster access to MRI. The hypothesis of the study is that a validated functional score would make it possible to sort the patients in the emergencies and to prescribe the MRI only in the cases of effective rupture of the LCA.

DETAILED DESCRIPTION:
A observational, Prospective, non-randomized, multi-centric study. The main objective of this study will be to determine the diagnostic performance (sensitivity and specificity) of a functional score for the detection of a rupture of the knee ACL in the immediate post-traumatic period.

It will follow the methodology for the evaluation of a new diagnostic test according to the STARD (Standards for Reporting of Diagnostic Accuracy) checklist.

Phases of the study

* Build score This phase will quantify the weight of each item and sub-items of the questionnaire already conceived from a statistical analysis adapted and thus to give a value to each item then a maximum value to the score.
* Validation of the score The score obtained will be validated in a different population versus MRI to determine its performance parameters. This score will be called the ACL-TS screening score (Tear Screening). An inter-evaluative reproducibility analysis of the score will be carried out in the investigative centers which have an emergency department
* Planned sample size For phase 1, a logistic regression will be performed. Empirically, there are 10 patients per variable for this questionnaire with 17 sub-items, 170 patients.

For Phase 2, the workforce was calculated on sensitivity because it is important to detect LCA ruptures. To obtain a sensitivity of 98% with a 2% CI, and taking into account a 10% rate of incomplete records, 210 patients should be included.

For the inter-evaluative ancillary reproducibility study, to obtain a Pearson coefficient of 0.8 (strong correlation if coefficient greater than 0.5) with a confidence interval of 0.67 to 0.88 and a risk of first 60 patients should be included.

Statistical analysis

* Analysis of normality of distributions
* Descriptive statistics: mean, standard deviation, minimum, maximum and median (quantitative variables); Frequency and percentage (qualitative variables).
* Comparisons of means: Student or Mann-Whitney according to the normality of the distributions
* Percentage comparisons: chi 2 or Fisher tests, idem
* The threshold of significance of the set of tests will be 0.05

Phase 1:

* A bi-varied study will then be carried out for each of the factors taken individually (search for an individual relationship, a rupture of the LCA confirmed by MRI vs the factors to be taken into account). These analyzes will provide an OR, an 95% CI of the OR, and a p-value measuring the severity of the association between the severe sprain and the factor taken into account.
* Follow a multivariate analysis (here logistic since the dependent variable will be "breaking ACL O / N"). To carry out this logistic regression, all factors for which p <0.25 will be included in the model. A descending step-by-step method will arrive at the final model which will contain only those factors whose p will be less than 5% and whose 95% CI of the OR will not contain 1. Possibly it will be possible to adjust The model on certain parameters and to look for possible interactions. The ORs and IC95% obtained will allow the gravity scores to be established.

Phase 2:

* Performance parameters of the score with respect to the MRI: ROC curves with determination of the optimal threshold value, calculation of the area under the curve (AUC), Se, Sp, the likelihood ratios positive and negative and the proportion of Subjects.
* Identify the factors that can modify the sensitivity of the score (age, sex, sport level, laxity, meniscal or cartilage lesions) by bi-varied analyzes between the group correctly classified by the MRI and the score And on the other hand the group presenting a discrepancy between the reference examination and the score. If several factors are identified, these analyzes may be supplemented by a multivariate logistic regression analysis
* Pearson correlation coefficient and intra-class correlation coefficient to evaluate all correlations between quantitative variables (score reproducibility, differential score / laxity)
* Model the diagnostic approach including the score by developing a decision tree

Inclusion procedure The study will target 380 patients seen in an emergency. After a knee sprain, patients usually go to hospital or a treatment center for medical consultation. For the study, patients will be recruited either in the emergency department if the investigating center has an emergency department or in the corresponding medical-surgical centers of the investigating center. Investigating surgeons at the centers should inform physicians of the initiation of the study and the modalities of implementation.

Usually, patients are received by an emergency physician, orthopedic surgeon on duty or a sports physician. A standard radiographic assessment will be performed to eliminate the presence of a bone fracture. If the patient meets the test selection criteria, he / she will be informed of the study and his / her right to oppose the collection of his / her medical data. The patient will ask all the questions necessary for his understanding before confirming his non-opposition. The questionnaire will then be completed by the physician with the patient. In the centers where the reproducibility study will be carried out, a second doctor will complete the questionnaire.

Once the consultation has been completed, the physician will issue prescriptions for the usual medical treatment, laximetry prescription (GNRB) to be performed between 3 to 6 weeks after the accident when the knee is indolent and the prescription of the MRI to be performed between 7 days and 1 month after the accident. The physician will inform the patient that they should consult with the investigator's orthopedic surgeon once the results of GNRB and MRI are available within 6 weeks of the accident.

During this delayed consultation, the orthopedic surgeon will realize in this patient the dynamic maneuvers of ligament testing. The study will end there for the patient. The surgeon will then follow his usual diagnostic procedure to decide on the future care of the patient.

Ethical aspects Agreement will be sought from the local Ethics committee. All patients will be fully informed and will be provided with an information form. The data will be entered into an internet page and will be analysed anonymously.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 55 years,
* Knee trauma occurred less than 9 days prior to hospital emergency visit or medical consultation,
* Absence of bone fractures on the standard radiographic assessment (face and profile),
* Patient affiliated to a social security scheme (beneficiary or beneficiary),
* Patient informed and confirmed his / her agreement to the study.

Exclusion Criteria:

* Severe knee trauma requiring immediate surgical management (fractures, dislocations)
* Traumatic history (including sprain) on the same or other knee
* Impossibility or refusal to do an MRI
* Inability to understand information delivered
* Patient's refusal
* Patients can not be tracked for geographical reasons

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will target patients seen in an emergency or hospital or a treatment center for medical consultation after a knee sprain.
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2017-04-29 (Actual); Primary Completion 2021-06-29 (Estimated); Study Completion 2021-08-29 (Estimated)

PRIMARY OUTCOMES:
Reference method or "gold standard" | Between 7 days and 2 months after the accident.
  MRI will be used to determine whether the LCA is broken. The direct signs of complete LCA rupture are based on its morphological study, signal and spatial orientation.
  * In the acute phase, haemarthrosis secondary to rupture appears as a T1-weighted hyposignal and a proton-density and T2 -weight hyper-signal. In the subacute phase, the proximal and distal stump retract and remain separated by a proton density and T2-weighted signaling area.
  * AND / OR: Horizontalisation of the ACL, evaluated in relation to the plane of the tibial plateaus or the Blumensaat line, indicates the complete character of the ACL rupture with a sensitivity of 89% and a specificity of 100%.
  * AND / OR: The "sign of the empty notch" to be sought in the frontal and axial planes is pathognomonic of the complete rupture of the LCA at its high insertion. It is the most frequent form of rupture

SECONDARY OUTCOMES:
Quantification of differential laxity with GNRB | Between 3 to 8 weeks after the accident
  The GNRB will be performed when the knee is indolent
Questionnaire of the score | At a day of patient inclusion
  This phase will quantify the weight of each item and sub-items of the questionnaire already conceived from a statistical analysis adapted and thus to give a value to each item then a maximum value to the score.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy NOURRISAT, PHD, Principal Investigator — Clinique des Maussins
Locations (1):
- Pr François-Xavier GUNEPIN, Lorient, France

IPD SHARING:
Plan to Share IPD: No
In this study, the individual participant data (IPD) is not available to other researchers

REFERENCES:
- [Background] Ahlden M, Hoshino Y, Samuelsson K, Araujo P, Musahl V, Karlsson J. Dynamic knee laxity measurement devices. Knee Surg Sports Traumatol Arthrosc. 2012 Apr;20(4):621-32. doi: 10.1007/s00167-011-1848-7. Epub 2011 Dec 31. PMID 22210516
- [Background] Bollen SR, Scott BW. Rupture of the anterior cruciate ligament--a quiet epidemic? Injury. 1996 Jul;27(6):407-9. doi: 10.1016/0020-1383(96)00033-2. PMID 8881137
- [Derived] Gunepin FX, Letartre R, Mouton C, Guillemot P, Common H, Thoreux P, Di Francia R, Graveleau N; Francophone Arthroscopy Society (SFA). Construction and validation of a functional diagnostic score in anterior cruciate ligament ruptures of the knee in the immediate post-traumatic period. Preliminary results of a multicenter prospective study. Orthop Traumatol Surg Res. 2023 Dec;109(8S):103686. doi: 10.1016/j.otsr.2023.103686. Epub 2023 Sep 28. PMID 37776951